CLINICAL TRIAL: NCT05619744
Title: An Open-Label, Multicenter Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Anti-Tumor Activity of RO7616789 in Participants With Advanced Small Cell Lung Cancer and Other Neuroendocrine Carcinomas
Brief Title: A Study to Evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Anti-tumor Activity of RO7616789 in Advanced Small Cell Lung Cancer and Other Neuroendocrine Carcinomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BP44382; 2023-506354-20-00 (Other: EU CT Number)
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Small Cell Lung Cancer; Neuroendocrine Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma, Neuroendocrine | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: RO7616789 QW: Dose Escalation (Experimental): Participants will receive a fixed dose of RO7616789 intravenously once weekly (QW) per dose level on Day 1, 8, and 15 of each 21-day cycle. In case of toxicity, step-up (single or double) dosing may be explored.
  Interventions: Drug: RO7616789; Drug: Tocilizumab
- Part 2: RO7616789 Q3W: Dose Escalation (Experimental): Participants will receive a fixed dose of RO7616789, at a dose determined in Part 1, intravenously once every 3 weeks (Q3W) on Day 1 of each 21-day cycle. In case of toxicity, step-up (single or double) dosing may be explored.
  Interventions: Drug: RO7616789; Drug: Tocilizumab
- Part 3: Dose Expansion (Experimental): Based on emerging data from Part 1 and 2, one or more dosing regimens will be further investigated in Part 3.
  Interventions: Drug: RO7616789; Drug: Tocilizumab

INTERVENTIONS:
Drug: RO7616789 — RO7616789 solution for infusion will be administered intravenously at a dose and per schedule as specified for the respective part.
Drug: Tocilizumab — Tocilizumab will be used as rescue therapy, in case of clinical presentation of cytokine release syndrome (CRS). Tocilizumab solution for infusion will be administered intravenously at 8 mg/kg for participants >/= 30 kg or at 12 mg/kg for participants < 30 kg.
  Other Names: Actemra, RoActemra

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and preliminary anti-tumor activity of RO7616789. The study will have 3 parts: Dose Escalation (Parts 1 and 2) and Dose Expansion (Part 3). Participants with advanced stage small cell lung cancer (SCLC) and neuroendocrine carcinoma (NEC) will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy at least 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate hematologic and end organ function
* Negative serum pregnancy test.
* Adequate contraception and no or interruption of breastfeeding
* Histologically confirmed extensive SCLC or poorly differentiated NEC of any other origin, relapsed after at least 1 systemic therapy
* Measurable disease according to Response Evaluation criteria in Solid Tumors (RECIST) Version 1.1
* Confirmed availability of representative archival tumor specimens in formalin-fixed, paraffin-embedded (FFPE) blocks or unstained slides

Exclusion Criteria:

* Pregnant or breastfeeding, or intending to become pregnant during the study or within 40 days after the final dose of study treatment
* Poorly controlled Type 2 diabetes mellitus defined as a screening hemoglobin A1c ≥ 8% or a fasting plasma glucose ≥ 160 mg/dL (or 8.8 mmol/L)
* QT interval corrected using Fridericia's formula (QTcF) > 470 ms. Abnormal electrocardiograms (ECGs) (triplicate) should be performed > 30 minutes apart
* Current treatment with medications that are well known to prolong the QT interval
* Prior treatment with anti-cluster of differentiation (CD)137 agents, anti-CD3 agents and/or delta-like ligand 3 (DLL3) targeted therapies
* Any anti-cancer therapy, whether investigational or approved, including chemotherapy, hormonal therapy, or radiotherapy, within 21 days prior to initiation of study treatment
* Any history of an immune-related Grade 4 adverse event (AE) attributed to prior anti-programmed death ligand-1 (PD-L1) /PD-1 or anti-cytotoxic T-lymphocyte-associated protein (CTLA-4) therapy (other than asymptomatic elevation of serum amylase or lipase)
* Any history of an immune-related Grade 3 adverse event attributed to prior anti-PD-L1 /PD-1 or anti-CTLA-4 therapy (other than asymptomatic elevation of serum amylase or lipase) that resulted in permanent discontinuation of the prior immunotherapeutic agent
* History or clinical evidence of primary central nervous system (CNS) malignancy, symptomatic CNS metastases, CNS metastases requiring any anti-tumor treatment, or leptomeningeal disease and current or history of CNS disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease
* Spinal cord compression that has not been definitively treated with surgery and/or radiation
* Active or history of clinically significant autoimmune disease
* Positive test for human immunodeficiency virus (HIV) infection
* Positive hepatitis B surface antigen (HbsAg) test, and/or positive total hepatitis B core antibody (HbcAb) test at screening
* Prior allogeneic hematopoietic stem cell transplantation or prior solid organ transplantation
* Administration of a live, attenuated vaccine within 4 weeks before first RO7616789 infusion
* Known allergy or hypersensitivity to any component of the RO7616789 formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-03-04 (Actual)

PRIMARY OUTCOMES:
Part 1, 2 and 3: Number of Participants with Adverse Events and Serious Adverse Events | Up to approximately 26 months
  Adverse events were reported according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0), and Cytokine release syndrome (CRS), will be graded based on the American Society for Transplantation and Cell Therapy (ASTCT) criteria.
Part 1 and 2: Number of Participants with Dose Limiting Toxicities (DLTs) | Day 1 through Day 21 in cycle 1 (Cycle is 21 days)
Part 3: Objective Response Rate (ORR) as determined by Investigator | Up to approximately 26 months
Part 3: Disease Control Rates as Determined by the Investigator | Up to approximately 26 months
Part 3: Duration of Response (DOR) as Determined by the Investigator | Up to approximately 26 months
Part 3: Progression Free Survival (PFS) as Determined by the Investigator | Up to approximately 26 months
Part 3: Overall Survival (OS) | Up to approximately 26 months

SECONDARY OUTCOMES:
Part 1, 2 and 3: Serum Concentration of RO7616789 | Up to approximately 26 months
Part 1, 2 and 3: Maximum Serum Concentration (Cmax) of RO7616789 | Up to approximately 26 months
Part 1, 2 and 3: Area Under the Concentration-Time Curve (AUC) of RO7616789 | Up to approximately 26 months
Part 1, 2 and 3: Total Clearance of RO7616789 | Up to approximately 26 months
Part 1, 2 and 3: Terminal Half-Life of RO7616789 | Up to approximately 26 months
Part 1, 2 and 3: Volume of Distribution of RO7616789 | Up to approximately 26 months
Part 1, 2 and 3: Time to Reach Steady State Concentration of RO7616789 | Up to approximately 26 months
Part 1, 2 and 3: Accumulation Ratio of RO7616789 | Up to approximately 26 months
Part 1 and 2: ORR as Determined by the Investigators | Up to approximately 26 months
Part 1 and 2: Disease Control Rates as Determined by the Investigator | Up to approximately 26 months
Part 1 and 2: DOR as Determined by the Investigators | Up to approximately 26 months
Part 1 and 2: PFS as Determined by the Investigators | Up to approximately 26 months
Part 1 and 2: OS as Determined by the Investigators | Up to approximately 26 months
Part 1, 2 and 3: Percentage of Participants With Anti-Drug Antibody (ADA) to RO7616789 | Up to approximately 26 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- United States (10):
  - Georgetown Uni Medical Center, Washington D.C., District of Columbia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - SCRI Oncology Partners, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Rigshospitalet, København Ø, Denmark
- Japan (2):
  - National Cancer Center Hospital East, Chiba
  - National Cancer Center Hospital, Tokyo
- Uniwersyteckie Centrum Kliniczne, Gda?sk, Poland
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing